CLINICAL TRIAL: NCT06490965
Title: Improving Obsessive-compulsive Disorder Treatments: from Lesions to Neuromodulation Targets
Acronym: ON-TARGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacao Champalimaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ON-TARGET; 31379 (Other Grant/Funding Number: 2023 NARSAD Young Investigator Grant, BBRF)
Record Dates: First submitted 2024-07-01; First posted 2024-07-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation; Neuronavigation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): Standard of care rTMS protocol, i.e., daily frequency of repetitive excitatory TMS at 20 Hz of the medial prefrontal cortex - approximate duration of each session between 40-60 minutes.
  Interventions: Other: Repetitive Transcranial Magnetic Stimulation; Other: Neuronavigation; Other: Magnetic Resonance Imaging
- Arm B (Experimental): Standard of care rTMS protocol, i.e., daily frequency of repetitive excitatory TMS at 20 Hz with adjustment of the stimulation site to primarily target the bilateral medial orbitofrontal cortex.
  Interventions: Other: Repetitive Transcranial Magnetic Stimulation; Other: Neuronavigation; Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Repetitive Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation (TMS) involves generating a magnetic field with specific spatial and temporal properties, allowing the induction of electric current in conductive material near this field. The electro-physiological principle of TMS is based on placing a coil over the skull that will induce a magnetic field generating action potentials in neuronal tissue in response to each TMS pulse. The repetitive application of TMS pulses (rTMS) allows for the modulation of neuronal excitability for a period after rTMS, ranging from inhibition, in the case of low frequencies (~1 Hz), or facilitation if high frequencies (equal to or greater than 5 Hz) are used.
  Other Names: rTMS; TMS; Non Invasive Brain Stimulation
Other: Neuronavigation — Neuronavigation is a non-invasive method that allows the creation of computerized three-dimensional models of brain structures based on neuroimaging exams of each individual (e.g., cranial magnetic resonance imaging). As such, this method has been used for various purposes, such as assisting in neurosurgery or mapping functional regions of the brain, but also in the context of TMS (Transcranial Magnetic Stimulation). In this latter area, its use as support for TMS has been employed for therapeutic, diagnostic, and research purposes. The neuronavigation system consists of several components, namely a locating camera, locators for the TMS coil, an adjustable headband with locators, a calibration system for these elements, and the neuronavigation software, which is installed on a supporting computer.
Other: Magnetic Resonance Imaging — Magnetic Resonance Imaging (MRI) is a non-invasive medical imaging technique that generates detailed images of the internal structures of the body using a strong magnetic field and radio waves. It provides high-resolution images of soft tissues, such as organs, muscles, and the brain, helping doctors diagnose and monitor various conditions, including injuries, tumors, and neurological disorders. MRI is particularly useful because it does not involve ionizing radiation, making it safer for patients than other imaging methods like X-rays or CT scans.
  Other Names: MRI

SUMMARY:
While in most cases of obsessive-compulsive disorder (OCD) a cause cannot be identified, this syndrome may develop as a consequence of focal brain lesions. Neuropsychiatric disorders secondary to brain insults are open windows to understand their underlying neurobiology. Different neuroimaging analysis methods, including pooled lesion topography and lesion network mapping, can be used to study lesional neuropsychiatric syndromes, including OCD. If successful, these strategies can also reveal new neuromodulation treatment targets, including for transcranial magnetic stimulation (TMS). Indeed, TMS targets to treat depression evolved from evidence extracted from lesional studies that were then refined and validated. For OCD treatment with TMS, already approved by the FDA and European Commission, targets were defined using a distinct approach, not involving causal brain lesions, which may contribute to lower than desirable remission rates. Lesional OCD is characterized by specific dysfunctional brain circuits. These circuits may be effectively targeted by TMS, which may optimize treatment of OCD. To address these hypotheses, we will test the therapeutic benefits of optimizing brain targets for the currently used TMS treatment of OCD, using information from the lesional-OCD brain network namely refining the target in the medial orbitofrontal cortex, bilaterally. Specifically, we will conduct a randomized clinical interventional study, using TMS to treat patients with OCD with inadequate response to other treatments, comparing, within the approved protocol for OCD treatment, the most frequently used stimulation site with a new target, adjusted according to the connectivity of lesions associated with the occurrence of OCD. If successful, our results may have immediate clinical implications in OCD treatment, as it will contribute to refine current therapeutic TMS strategies for OCD and defining new clinical research strategies in this domain.

DETAILED DESCRIPTION:
In this study, we hypothesize that the cortical region identified from connectivity networks associated with lesional OCD may be a more effective TMS stimulation site than the one currently used in OCD treatment. Thus, we intend to compare the efficacy of the TMS protocol as approved for OCD, between its application at the currently used stimulation site (bilateral dorsomedial prefrontal cortex) and its application at an adjusted stimulation site, according to the more specific cortical areas of dysfunctional circuits associated with lesional OCD, namely the bilateral medial orbitofrontal cortex (OFC) region.

The participants in this study will be recruited at the Champalimaud Foundation. The physicians on the research team will identify patients who are being treated for OCD in the Neuropsychiatry Unit, or who are referred to the unit for this purpose. In this study, we aim to prospectively recruit 32 individuals according to the eligibility criteria specified in the respective section.

We propose to conduct a randomized, double-blinded interventional study, open only to the technician administering the treatment. After agreeing to participate in the study, the participant will be invited to attend the first study visit. There, participants will be assigned a unique identification number to maintain their anonymity in the study. Then, a qualified team member will ask the participant to complete the sociodemographic and clinical questionnaire to confirm the conditions for TMS and MRI, including an appropriate screening tool for the occurrence of seizures and/or epilepsy. The Mini International Neuropsychiatric Interview (MINI) and he Structured Clinical Interview for Diagnostic and statistical manual of mental disorders (SCID) will serve the purpose of verifying the eligibility criteria of the study participant, including confirmation of the OCD diagnosis, using SCID. After confirming their eligibility, the participant will be invited to complete the remaining psychometric assessment, which will reflect the baseline values of each instrument. The following will be assessed: YBOCS-II (primary outcome), BDI-II, OCI-R, STAI, World Health Organization Five Well-Being Index (WHO-5), and YMRS (secondary outcomes), and Edinburgh Handedness Inventory (EHI).

In this study, to ensure that the TMS target site used is precisely located, we will use neuronavigation in each TMS session performed. Thus, in the next step of the first visit, the participant will be invited to undergo an MRI scan. This procedure cannot be waived, as without the MRI scan of each individual, the appropriate use of neuronavigation is compromised. If the participant cannot or does not want to undergo this procedure, they will be excluded from the study. The MRI protocol will include the collection of structural and functional neuroimaging data. The duration of this neuroimaging exam will be approximately 20-30 minutes.

After completing this step, the participant will be randomized to one of the two study arms. Please see details of each study arm in the respective section. The first visit of the TMS treatment cycle will be scheduled later. During this first visit of the TMS treatment cycle, the motor hotspot and the motor excitability threshold will be determined, which will be subsequently used to define the appropriate treatment intensity for each individual. Finally, the stimulation site will be determined using the neuronavigation system utilizing each individual's MRI scan. It is emphasized that the stimulation site will be mandatory determined at all TMS treatment visits. The TMS protocol will then commence, characterized by 20 Hz frequency irrespective of study arm. At the beginning of each TMS treatment cycle visit, the presence of potential side effects since the last TMS session will be screened. Every 5 TMS treatment cycle visits (1st, 6th, 11th, 16th, 21st, and 26th visits), the following psychometric scales will be repeated at the beginning of each visit: BDI-II, WHO-5, OCI-R, and YMRS (secondary outcomes). Every 5 TMS treatment cycle visits (1st, 6th, 11th, 16th, 21st, and 26th visits), the motor hotspot and the motor excitability threshold will be redefined, and consequently, the treatment stimulation intensity will be adjusted. At the end of each TMS treatment cycle visit, the next visit will be scheduled to occur on a daily basis, on business days, for a total of 30 visits. After the end of the TMS treatment cycle, the last study visit will be scheduled (primary endpoint, end-of-study visit), which should preferably occur between 2-3 weeks after the 30th TMS treatment cycle visit. During this visit, the YBOCS-II (primary outcome) will be applied. Participants will also be invited to undergo a new MRI scan, with the same characteristics as identified above.

Clinical efficacy will be assessed by changes in the severity of OCD symptoms compared to baseline, evaluated (using YBOCS-II; primary outcome) after 30 daily sessions of TMS, comparing the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years;
* Established diagnosis of Obsessive-Compulsive Disorder according to Diagnostic and statistical manual of mental disorders 5 (DSM5) criteria;
* Capacity to give consent;
* Fluent in Portuguese and/or English;
* If potential for pregnancy, agrees to use an effective method of contraception throughout the study period.

Exclusion Criteria:

* Obsessive-compulsive symptoms severity assessed at baseline visit with the instrument Yale-Brown Obsessive Compulsive Scale - II (YBOCS-II) ≤ 24;
* Presence of uncontrolled active medical illness;
* Known structural lesion of the central nervous system;
* Electric or metallic implants in the body not compatible with electromagnetic radiation;
* Electric or metallic brain implants;
* Cardiac implants;
* Epilepsy;
* Pregnant, breastfeeding, or planning pregnancy women;
* Alcohol or substance abuse and/or dependence;
* Major Neurocognitive Disorder;
* Developmental disorders with low intelligence quotient or any other form of cognitive deficit;
* Active neurological disease;
* Individuals presenting with any psychotic or mood disorder requiring hospitalization at the time of eligibility criteria assessment;
* Contraindication for performing MRI;
* Individuals who have already been treated for OCD with TMS;
* Any other reason that renders the individual unable to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale - II (YBOCS-II) | Before and after TMS treatment cycle. The latter will be considered the primary endpoint (end-of-study visit) and will occur preferably between 2-3 weeks after last TMS session.
  Assessment instrument for the severity of OCD symptoms; scores can range from 0-50; higher scores mean worse outcome.

SECONDARY OUTCOMES:
State Trait Anxiety Inventory (STAI) | Before and after TMS treatment cycle. The latter will be considered the primary endpoint (end-of-study visit) and will occur preferably between 2-3 weeks after last TMS session.
  Self-report instrument that measures anxiety in the dimensions of state anxiety and trait anxiety that often occur in comorbidity with OCD symptoms; scores for both state anxiety and trait anxiety can range from 20-80; higher scores mean worse outcome for both state anxiety and trait anxiety.
Beck Depression Inventory II (BDI-II) | Before TMS treatment cycle. Every 5 TMS treatment cycle visits (1st, 6th, 11th, 16th, 21st, and 26th visits). After TMS treatment cycle, i.e., 2-3 weeks after last TMS session.
  Self-report scale that measures the severity of depressive symptoms often occurring in comorbidity with OCD symptoms; scores can range from 0-63; higher scores mean worse outcome.
Obsessive-Compulsive Inventory - Revised (OCI-R) | Before TMS treatment cycle. Every 5 TMS treatment cycle visits (1st, 6th, 11th, 16th, 21st, and 26th visits). After TMS treatment cycle, i.e., 2-3 weeks after last TMS session.
  Self-report scale that allows the assessment of dimensions present in OCD; scores can range from 0-72; higher scores mean worse outcome.
Young Mania Rating Scale (YMRS) | Before TMS treatment cycle. Every 5 TMS treatment cycle visits (1st, 6th, 11th, 16th, 21st, and 26th visits). After TMS treatment cycle, i.e., 2-3 weeks after last TMS session.
  Assessment instrument for the severity of manic symptoms, a possible neuropsychiatric adverse effect of TMS; scores can range from 0-60; higher scores mean worse outcome.
World Health Organization Five Well-Being Index (WHO-5) | Before TMS treatment cycle. Every 5 TMS treatment cycle visits (1st, 6th, 11th, 16th, 21st, and 26th visits). After TMS treatment cycle, i.e., 2-3 weeks after last TMS session.
  Self-report scale that measures subjective quality of life based on mood, vitality, and interest in things in general; scores can range from 0-25; higher scores mean better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gonçalo Cotovio, MD, PhD, Principal Investigator — Champalimaud Foundation; Albino J. Oliveira-Maia, MD, MPH, PhD, Principal Investigator — Champalimaud Foundation
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
To date there is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Ondrako JM, Ornston LN. Biological distribution and physiological role of the beta-ketoadipate transport system. J Gen Microbiol. 1980 Sep;120(1):199-209. doi: 10.1099/00221287-120-1-199. PMID 7217919
- [Background] Carmi L, Alyagon U, Barnea-Ygael N, Zohar J, Dar R, Zangen A. Clinical and electrophysiological outcomes of deep TMS over the medial prefrontal and anterior cingulate cortices in OCD patients. Brain Stimul. 2018 Jan-Feb;11(1):158-165. doi: 10.1016/j.brs.2017.09.004. Epub 2017 Sep 6. PMID 28927961
- [Background] Carmi L, Tendler A, Bystritsky A, Hollander E, Blumberger DM, Daskalakis J, Ward H, Lapidus K, Goodman W, Casuto L, Feifel D, Barnea-Ygael N, Roth Y, Zangen A, Zohar J. Efficacy and Safety of Deep Transcranial Magnetic Stimulation for Obsessive-Compulsive Disorder: A Prospective Multicenter Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):931-938. doi: 10.1176/appi.ajp.2019.18101180. Epub 2019 May 21. PMID 31109199
- [Background] Cocchi L, Naze S, Robinson C, Webb L, Sonkusare S, Hearne LJ, et al. Effects of transcranial magnetic stimulation of the rostromedial prefrontal cortex in obsessive-compulsive disorder: a randomized clinical trial. Nat Mental Health. 2023 Jul 24;1(8):555-63.
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Cook DA, Beckman TJ. Current concepts in validity and reliability for psychometric instruments: theory and application. Am J Med. 2006 Feb;119(2):166.e7-16. doi: 10.1016/j.amjmed.2005.10.036. PMID 16443422
- [Background] Cotovio G, Talmasov D, Barahona-Correa JB, Hsu J, Senova S, Ribeiro R, Soussand L, Velosa A, Silva VCE, Rost N, Wu O, Cohen AL, Oliveira-Maia AJ, Fox MD. Mapping mania symptoms based on focal brain damage. J Clin Invest. 2020 Oct 1;130(10):5209-5222. doi: 10.1172/JCI136096. PMID 32831292
- [Background] Cotovio G, Ventura F, Rodrigues da Silva D, Pereira P, Oliveira-Maia AJ. Regulatory Clearance and Approval of Therapeutic Protocols of Transcranial Magnetic Stimulation for Psychiatric Disorders. Brain Sci. 2023 Jul 5;13(7):1029. doi: 10.3390/brainsci13071029. PMID 37508962
- [Background] Feffer K, Fettes P, Giacobbe P, Daskalakis ZJ, Blumberger DM, Downar J. 1Hz rTMS of the right orbitofrontal cortex for major depression: Safety, tolerability and clinical outcomes. Eur Neuropsychopharmacol. 2018 Jan;28(1):109-117. doi: 10.1016/j.euroneuro.2017.11.011. Epub 2017 Nov 17. PMID 29153927
- [Background] Fitzgerald, Paul B., and Z. Jeff Daskalakis. Repetitive Transcranial Magnetic Stimulation Treatment for Depressive Disorders: A Practical Guide. Heidelberg: Springer, 2013.
- [Background] Fitzsimmons SMDD, van der Werf YD, van Campen AD, Arns M, Sack AT, Hoogendoorn AW; other members of the TETRO Consortium; van den Heuvel OA. Repetitive transcranial magnetic stimulation for obsessive-compulsive disorder: A systematic review and pairwise/network meta-analysis. J Affect Disord. 2022 Apr 1;302:302-312. doi: 10.1016/j.jad.2022.01.048. Epub 2022 Jan 15. PMID 35041869
- [Background] Herwig U, Padberg F, Unger J, Spitzer M, Schonfeldt-Lecuona C. Transcranial magnetic stimulation in therapy studies: examination of the reliability of "standard" coil positioning by neuronavigation. Biol Psychiatry. 2001 Jul 1;50(1):58-61. doi: 10.1016/s0006-3223(01)01153-2. PMID 11457424
- [Background] Herwig U, Schonfeldt-Lecuona C, Wunderlich AP, von Tiesenhausen C, Thielscher A, Walter H, Spitzer M. The navigation of transcranial magnetic stimulation. Psychiatry Res. 2001 Nov 30;108(2):123-31. doi: 10.1016/s0925-4927(01)00121-4. PMID 11738546
- [Background] Horn A, Reich M, Vorwerk J, Li N, Wenzel G, Fang Q, Schmitz-Hubsch T, Nickl R, Kupsch A, Volkmann J, Kuhn AA, Fox MD. Connectivity Predicts deep brain stimulation outcome in Parkinson disease. Ann Neurol. 2017 Jul;82(1):67-78. doi: 10.1002/ana.24974. PMID 28586141
- [Background] Ikawa H, Osawa R, Sato A, Mizuno H, Noda Y. A Case Series of Deep Transcranial Magnetic Stimulation Treatment for Patients with Obsessive-Compulsive Disorder in the Tokyo Metropolitan Area. J Clin Med. 2022 Oct 18;11(20):6133. doi: 10.3390/jcm11206133. PMID 36294453
- [Background] Jahanshahi M, Ridding MC, Limousin P, Profice P, Fogel W, Dressler D, Fuller R, Brown RG, Brown P, Rothwell JC. Rapid rate transcranial magnetic stimulation--a safety study. Electroencephalogr Clin Neurophysiol. 1997 Dec;105(6):422-9. doi: 10.1016/s0924-980x(97)00057-x. PMID 9448643
- [Background] Johnson KA, Baig M, Ramsey D, Lisanby SH, Avery D, McDonald WM, Li X, Bernhardt ER, Haynor DR, Holtzheimer PE 3rd, Sackeim HA, George MS, Nahas Z. Prefrontal rTMS for treating depression: location and intensity results from the OPT-TMS multi-site clinical trial. Brain Stimul. 2013 Mar;6(2):108-17. doi: 10.1016/j.brs.2012.02.003. Epub 2012 Mar 14. PMID 22465743
- [Background] Khedr EM, Elbeh K, Saber M, Abdelrady Z, Abdelwarith A. A double blind randomized clinical trial of the effectiveness of low frequency rTMS over right DLPFC or OFC for treatment of obsessive-compulsive disorder. J Psychiatr Res. 2022 Dec;156:122-131. doi: 10.1016/j.jpsychires.2022.10.025. Epub 2022 Oct 10. PMID 36244200
- [Background] Kupfer DJ, Frank E, Phillips ML. Major depressive disorder: new clinical, neurobiological, and treatment perspectives. Lancet. 2012 Mar 17;379(9820):1045-55. doi: 10.1016/S0140-6736(11)60602-8. Epub 2011 Dec 19. PMID 22189047
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Loo CK, McFarquhar TF, Mitchell PB. A review of the safety of repetitive transcranial magnetic stimulation as a clinical treatment for depression. Int J Neuropsychopharmacol. 2008 Feb;11(1):131-47. doi: 10.1017/S1461145707007717. Epub 2007 Sep 20. PMID 17880752
- [Background] Machii K, Cohen D, Ramos-Estebanez C, Pascual-Leone A. Safety of rTMS to non-motor cortical areas in healthy participants and patients. Clin Neurophysiol. 2006 Feb;117(2):455-71. doi: 10.1016/j.clinph.2005.10.014. Epub 2006 Jan 4. PMID 16387549
- [Background] Maia TV, Cooney RE, Peterson BS. The neural bases of obsessive-compulsive disorder in children and adults. Dev Psychopathol. 2008 Fall;20(4):1251-83. doi: 10.1017/S0954579408000606. PMID 18838041
- [Background] Mayberg HS, Liotti M, Brannan SK, McGinnis S, Mahurin RK, Jerabek PA, Silva JA, Tekell JL, Martin CC, Lancaster JL, Fox PT. Reciprocal limbic-cortical function and negative mood: converging PET findings in depression and normal sadness. Am J Psychiatry. 1999 May;156(5):675-82. doi: 10.1176/ajp.156.5.675. PMID 10327898
- [Background] McClintock SM, Reti IM, Carpenter LL, McDonald WM, Dubin M, Taylor SF, Cook IA, O'Reardon J, Husain MM, Wall C, Krystal AD, Sampson SM, Morales O, Nelson BG, Latoussakis V, George MS, Lisanby SH; National Network of Depression Centers rTMS Task Group; American Psychiatric Association Council on Research Task Force on Novel Biomarkers and Treatments. Consensus Recommendations for the Clinical Application of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Depression. J Clin Psychiatry. 2018 Jan/Feb;79(1):16cs10905. doi: 10.4088/JCP.16cs10905. PMID 28541649
- [Background] Mutz J, Edgcumbe DR, Brunoni AR, Fu CHY. Efficacy and acceptability of non-invasive brain stimulation for the treatment of adult unipolar and bipolar depression: A systematic review and meta-analysis of randomised sham-controlled trials. Neurosci Biobehav Rev. 2018 Sep;92:291-303. doi: 10.1016/j.neubiorev.2018.05.015. Epub 2018 May 12. PMID 29763711
- [Background] Nauczyciel C, Le Jeune F, Naudet F, Douabin S, Esquevin A, Verin M, Dondaine T, Robert G, Drapier D, Millet B. Repetitive transcranial magnetic stimulation over the orbitofrontal cortex for obsessive-compulsive disorder: a double-blind, crossover study. Transl Psychiatry. 2014 Sep 9;4(9):e436. doi: 10.1038/tp.2014.62. PMID 25203167
- [Background] Council for International Organizations of Medical Sciences. International ethical guidelines for biomedical research involving human subjects. Bull Med Ethics. 2002 Oct;(182):17-23. PMID 14983848
- [Background] Perera T, George MS, Grammer G, Janicak PG, Pascual-Leone A, Wirecki TS. The Clinical TMS Society Consensus Review and Treatment Recommendations for TMS Therapy for Major Depressive Disorder. Brain Stimul. 2016 May-Jun;9(3):336-346. doi: 10.1016/j.brs.2016.03.010. Epub 2016 Mar 16. PMID 27090022
- [Background] Radhu N, de Jesus DR, Ravindran LN, Zanjani A, Fitzgerald PB, Daskalakis ZJ. A meta-analysis of cortical inhibition and excitability using transcranial magnetic stimulation in psychiatric disorders. Clin Neurophysiol. 2013 Jul;124(7):1309-20. doi: 10.1016/j.clinph.2013.01.014. Epub 2013 Feb 26. PMID 23485366
- [Background] Rehn S, Eslick GD, Brakoulias V. A Meta-Analysis of the Effectiveness of Different Cortical Targets Used in Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Obsessive-Compulsive Disorder (OCD). Psychiatr Q. 2018 Sep;89(3):645-665. doi: 10.1007/s11126-018-9566-7. PMID 29423665
- [Background] Robinson RG, Starkstein SE. Mood disorders following stroke: new findings and future directions. J Geriatr Psychiatry. 1989;22(1):1-15. PMID 2607085
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Roth Y, Tendler A, Arikan MK, Vidrine R, Kent D, Muir O, MacMillan C, Casuto L, Grammer G, Sauve W, Tolin K, Harvey S, Borst M, Rifkin R, Sheth M, Cornejo B, Rodriguez R, Shakir S, Porter T, Kim D, Peterson B, Swofford J, Roe B, Sinclair R, Harmelech T, Zangen A. Real-world efficacy of deep TMS for obsessive-compulsive disorder: Post-marketing data collected from twenty-two clinical sites. J Psychiatr Res. 2021 May;137:667-672. doi: 10.1016/j.jpsychires.2020.11.009. Epub 2020 Nov 4. PMID 33183769
- [Background] Ruffini C, Locatelli M, Lucca A, Benedetti F, Insacco C, Smeraldi E. Augmentation effect of repetitive transcranial magnetic stimulation over the orbitofrontal cortex in drug-resistant obsessive-compulsive disorder patients: a controlled investigation. Prim Care Companion J Clin Psychiatry. 2009;11(5):226-30. doi: 10.4088/PCC.08m00663. PMID 19956460
- [Background] Seybert C, Cotovio G, Rodrigues da Silva D, Faro Viana F, Pereira P, Oliveira-Maia AJ. Replicability of motor cortex-excitability modulation by intermittent theta burst stimulation. Clin Neurophysiol. 2023 Aug;152:22-33. doi: 10.1016/j.clinph.2023.04.014. Epub 2023 May 18. PMID 37269770
- [Background] Siddiqi SH, Schaper FLWVJ, Horn A, Hsu J, Padmanabhan JL, Brodtmann A, Cash RFH, Corbetta M, Choi KS, Dougherty DD, Egorova N, Fitzgerald PB, George MS, Gozzi SA, Irmen F, Kuhn AA, Johnson KA, Naidech AM, Pascual-Leone A, Phan TG, Rouhl RPW, Taylor SF, Voss JL, Zalesky A, Grafman JH, Mayberg HS, Fox MD. Brain stimulation and brain lesions converge on common causal circuits in neuropsychiatric disease. Nat Hum Behav. 2021 Dec;5(12):1707-1716. doi: 10.1038/s41562-021-01161-1. Epub 2021 Jul 8. PMID 34239076
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835
- [Background] Spampinato C, Aguglia E, Concerto C, Pennisi M, Lanza G, Bella R, Cantone M, Pennisi G, Kavasidis I, Giordano D. Transcranial magnetic stimulation in the assessment of motor cortex excitability and treatment of drug-resistant major depression. IEEE Trans Neural Syst Rehabil Eng. 2013 May;21(3):391-403. doi: 10.1109/TNSRE.2013.2256432. Epub 2013 Apr 3. PMID 23559064
- [Background] Trapp NT, Bruss J, King Johnson M, Uitermarkt BD, Garrett L, Heinzerling A, Wu C, Koscik TR, Ten Eyck P, Boes AD. Reliability of targeting methods in TMS for depression: Beam F3 vs. 5.5 cm. Brain Stimul. 2020 May-Jun;13(3):578-581. doi: 10.1016/j.brs.2020.01.010. Epub 2020 Jan 14. PMID 32289680
- [Background] Tzirini M, Roth Y, Harmelech T, Zibman S, Pell GS, Kimiskidis VK, Tendler A, Zangen A, Samaras T. Detailed measurements and simulations of electric field distribution of two TMS coils cleared for obsessive compulsive disorder in the brain and in specific regions associated with OCD. PLoS One. 2022 Aug 30;17(8):e0263145. doi: 10.1371/journal.pone.0263145. eCollection 2022. PMID 36040972
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Weigand A, Horn A, Caballero R, Cooke D, Stern AP, Taylor SF, Press D, Pascual-Leone A, Fox MD. Prospective Validation That Subgenual Connectivity Predicts Antidepressant Efficacy of Transcranial Magnetic Stimulation Sites. Biol Psychiatry. 2018 Jul 1;84(1):28-37. doi: 10.1016/j.biopsych.2017.10.028. Epub 2017 Nov 10. PMID 29274805